CLINICAL TRIAL: NCT02268799
Title: High Sensitivity Troponin T Levels Following Elective External Direct Current Cardioversion for Atrial Fibrillation / Atrial Flutter
Brief Title: High Sensitivity Troponin T Levels Following DC Cardioversion for Atrial Fibrillation / Atrial Flutter
Status: Completed | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Ronstan Lobo, MB, BMedSc, MRCPI, MRCP(UK), Dr., University of Limerick
Other Study IDs: RL002
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Cardioversion; High Sensitivity Troponin T (Hs-Trop T); Brain Natriuretic Peptide (BNP); Neutrophil Gelatinase-associated Lipocalin (NGAL)
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DC Cardioversion: Patients undergoing DC cardioversion

SUMMARY:
The purpose of this study is to determine if there is a rise in serum high sensitivity troponin T (a marker for heart muscle injury) following a direct current cardioversion (shock therapy) used for patients with atrial fibrillation. This will help us determine if direct current cardioversion results in damage to the heart muscles in a sufficient amount to cause a rise in high sensitivity troponin T.

DETAILED DESCRIPTION:
High sensitivity Troponin T is a relatively new biomarker that is highly sensitive and specific for myocardial injury. Its widespread use has helped in the determination and investigation for myocardial ischemia in patients. Previous studies have shown a rise in creatine kinase (CK) and the more specific creatine kinase-MB isoenzyme (CKMB) after DC cardioversion. Studies on the earlier generation troponin T found that the levels don't rise or rise only minimally after DC cardioversion. The high sensitivity troponin T has never been studied in the setting of DC cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation / atrial flutter attending for direct current external cardioversion
* Age 18 or older

Exclusion Criteria:

* Myocardial infarction within the last 6 weeks
* Coronary artery bypass grafting, percutaneous coronary intervention or any other invasive cardiac procedure within the last 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation/flutter who attend the Coronary Care Unit of the University Hospital Limerick for a pre-organised appointment for direct current external cardioversion will be requested to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
High Sensitivity Troponin T levels pre and 6 hours post cardioversion | 1 year

SECONDARY OUTCOMES:
Creatine Kinase levels pre and 6 hours post cardioversion | 1 year
B-type Natriuretic Peptide (BNP) levels pre and 6 hours post cardioversion | 1 year
Neutrophil Gelatinase-associated Lipocalin (NGAL) levels pre and 6 hours post cardioversion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kiernan, MD, Study Chair — University of Limerick
Locations (1):
- University Hospital Limerick, Dooradoyle, Limerick, Ireland